CLINICAL TRIAL: NCT05060172
Title: A Cross-sectional, Interventional, Single-arm Clinical Study for Validating the Equivalence of Bloomlife MFM-Pro to Clinical Standard-of-care for Antepartum Fetal Monitoring
Brief Title: A Clinical Study for Validating the Equivalence of Bloomlife MFM-Pro to Clinical Standard-of-care for Antepartum Fetal Monitoring
Acronym: NST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bloom Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NST-01-2020-EU
Record Dates: First submitted 2021-05-31; First posted 2021-09-29 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Fetal Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bloomlife MFM-Pro (Experimental)
  Interventions: Device: Bloomlife MFM-Pro

INTERVENTIONS:
Device: Bloomlife MFM-Pro — Bloomlife MFM-Pro is a non-invasive, wireless, external monitoring system used to measure fetal heart rate, maternal heart rate, and uterine activity during antepartum (non-stress) testing on pregnant women with a singleton pregnancy.
  The system acquires biopotential signals from abdominal surface electrodes and measures the fetal electrocardiography, maternal electrocardiography, electrohysterography, as well as accelerometer data.

SUMMARY:
Bloomlife has developed a wearable system (Bloomlife MFM-Pro) that can allow fetal monitoring to be conveniently performed in healthcare settings under supervision of a healthcare professional.

Bloomlife MFM-Pro is a non-invasive, wireless, external monitoring system used to measure fetal heart rate, maternal heart rate, and uterine activity during antepartum (non-stress) testing on pregnant women with a singleton pregnancy.

The purpose of this study is to validate that the Bloomlife MFM-Pro is equivalent to clinical standard-of-care for routine non-stress test (NST) performed at the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman ≥ 18 years old
* Gestational age ≥ 32 weeks and 0 days
* Singleton pregnancy
* Ability to read and understand Dutch or English
* Willingness to participate in the study

Exclusion Criteria:

* Implanted pacemaker or any other implanted electrical device
* Plurality higher than 1
* History of allergies to skin adhesives
* Contraindication to the use of the CTG

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Extent of agreement between Bloomlife MFM-Pro and CTG in fetal heart rate | 1 hour
  Bland-Altman analysis, based on a 95% limits of agreement
Extent of agreement between Bloomlife MFM-Pro and CTG in maternal heart rate | 1 hour
  Bland-Altman analysis, based on a 95% limits of agreement

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Gyselaers, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided